CLINICAL TRIAL: NCT01008176
Title: Restoring Sleep Homeostasis to Lower Blood Pressure: A Behavioral Prevention and Treatment Approach
Brief Title: Restoring Sleep Homeostasis to Lower Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Monika Haack, Assistant Professor of Neurology, Beth Israel Deaconess Medical Center
Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2005P000246
Record Dates: First submitted 2009-10-20; First posted 2009-11-05 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Hypertension; Pre-hypertension
Keywords: Hypertension; Sleep; Blood Pressure; Inflammatory Markers
MeSH Terms: conditions — Hypertension; Prehypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Sleep extension — Habitual sleep duration is extended by 60min/night over a 6-week time period.

SUMMARY:
Cutting back on sleep duration has developed into a common, highly prevalent habit in the adult population, and may lead to a major health problem. Large epidemiological studies have demonstrated that short sleep duration is associated with increased risk of cardiovascular disease (CVD). The investigators' preliminary data on the effects of experimental sleep reduction have shown elevation of blood pressure (BP) and inflammatory markers, such as interleukin-6 (IL-6) and C reactive protein (CRP), suggesting that both may play an important role in linking sleep loss and CVD risk. With this background, the investigators hypothesize that restoring sleep homeostasis, i. e. getting adequate amounts of sleep, is an effective behavioral intervention in the treatment of elevated BP.

The investigators will test this hypothesis in subjects with BP above normal and with short habitual sleep duration, as verified by sleep logs and actigraphic recordings. Subjects will either undergo 6 weeks of mild sleep extension, in which 60 min of bedtime will be added to the habitual sleep duration, or subjects will maintain their habitual sleep duration for the following 6 weeks.

Regarding their first specific aim, the investigators expect that sleep extension across 6 weeks will lower BP, inflammatory (IL-6, CRP, cell adhesion molecules) and autonomic markers (catecholamines). In particular, the investigators expect that in subjects with mild BP elevation, i. e. with pre-hypertension, sleep extension leads to normalization of BP.

This study presents a very first approach in using sleep behavior components for the treatment of elevated BP. Therefore, the investigators' second specific aim will characterize the strength of associations between changes in sleep duration, BP, and inflammation, and they will explore factors that are predictive for these changes. In particular, adiposity, as measured by percent body fat, has frequently been shown to be related to short sleep duration and inflammatory processes, but the role of adiposity in modulating the physiological consequences of changes in sleep duration has never been addressed.

If the investigators' hypothesis is correct, sleep extension may be considered as an additional component in current lifestyle intervention programs in combating and preventing hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Current history of prehypertension or stage 1 hypertension
* Sleep duration <= 7 hours/night

Exclusion Criteria:

* Sleep disorders
* History of psychiatric or severe medical disorders
* regular medication intake, except anti-hypertensive and birth control medication

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2005-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure | 6 weeks

SECONDARY OUTCOMES:
Change in inflammatory and autonomic markers (IL-6, CRP, norepinephrine) | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: haack monika, md, Principal Investigator — doctor
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Haack M, Serrador J, Cohen D, Simpson N, Meier-Ewert H, Mullington JM. Increasing sleep duration to lower beat-to-beat blood pressure: a pilot study. J Sleep Res. 2013 Jun;22(3):295-304. doi: 10.1111/jsr.12011. Epub 2012 Nov 22. PMID 23171375